CLINICAL TRIAL: NCT00843778
Title: A Phase IIIB, Multi-center, Open Label Follow-up Study to Evaluate the Safety and Efficacy of Certolizumab Pegol Administered Concomitantly With DMARDs in Patients With Active Rheumatoid Arthritis Who Participated in C87076.
Brief Title: Follow-up of Rheumatoid Arthritis (RA) Moderate to Low Disease Activity Study
Acronym: CERTAIN 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87080; 2007-000830-38 (EudraCT Number)
Record Dates: First submitted 2009-01-05; First posted 2009-02-13 (Estimated); Results first posted 2013-10-31 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Moderate to Low Disease Activity; Certolizumab Pegol
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab Pegol (Experimental): Certolizumab Pegol 200 mg every two weeks at the hospital by a nurse. Certolizumab Pegol 200 mg every two weeks at the patient's home done by patient (self-injection).
  Interventions: Biological: Certolizumab Pegol

INTERVENTIONS:
Biological: Certolizumab Pegol — 200 mg every two weeks
  Certolizuimab Pegol 200 mg every two weeks Subjects who flared at Week 48 or Week 52 of feeder study C87076 [NCT00674362], will receive respectively once 400 mg Certolizumab Pegol or three times 400 mg Certolizumab Pegol at two weeks interval as part of an induction phase in the C87080 study. Thereafter the subject enters the C87080 study and will be further treated with 200 mg Certolizumab Pegol every two weeks.
  Other Names: Cimzia; CDP870

SUMMARY:
To continue to assess the clinical safety and efficacy of Certolizumab Pegol as add-on therapy with stable-dose Disease Modifying Anti-Rheumatic Drugs (DMARDs)

DETAILED DESCRIPTION:
This is a Phase IIIB, multi-centre, open-label, follow-up study to study C87076 [NCT00674362] designed to continue to assess the safety and efficacy of Certolizumab Pegol.

Two different population will enter the study from C87076 [NCT00674362] and will be treated with Certolizumab Pegol every two weeks until it is commercially available for the indication of Rheumatoid Arthritis (RA) in the subject's country or region or until further notice from UCB:

Population 1: Are those subjects who failed to achieve remission at Week 20 and/or Week 24 and who completed the Week 24 assessment of study C86076 [NCT00674362].The Week 24 assessment (visit 14) of C87076 [NCT00674362] will also be the entry assessment (visit 1) for C87080. The subjects will receive Certolizumab Pegol 200 mg every two weeks. No induction period will be applied to ensure the blinding of study C87076 [NCT00674362].

Population 2: Are those subjects who achieved remission at both Week 20 and Week 24, flared up between Week 24 and Week 52 and completed the Week 52 assessment in study C87076 [NCT00674362]. The Week 52 assessment (visit 26) of C87076 [NCT00674362] will also be the entry assessment (visit 1) for C87080.

Subjects who flared prior to Week 48 in the C87076 [NCT00674362] study will receive Certolizumab Pegol 200 mg every two weeks in the C87080 study.

Those who flared at Week 48 or Week 52, will receive respectively once 400 mg Certolizumab Pegol or three times 400 mg Certolizumab Pegol at two weeks interval as part of an induction phase in the C87080 study. Thereafter the subject enters the C87080 study and will be further treated with 200 mg Certolizumab Pegol every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established adult rheumatoid arthritis on Disease Modifying Anti-Rheumatic Drugs (DMARDs) therapy who were included in C87076 protocol and:
* either failed to achieve remission after 6 months of study treatment
* or flared after the 6 months of study treatment and completed the study (C87076 [NCT00674362])

Exclusion Criteria:

* All the concomitant diseases or pathological conditions that could interfere and impact the assessment of the study treatment
* Previous clinical trials and previous biological therapy that could interfere with the results in the present clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (25):
- 6, Vienna, Austria
- France (3):
  - 11, Rennes
  - 64, Toulouse
  - 10, Tours
- Germany (10):
  - 17, Berlin
  - 47, Berlin
  - 20, Erlangen
  - 50, Essen
  - 16, Frankfurt
  - 19, Heidelberg
  - 15, Herne
  - 24, Ratingen
  - 18, Vogelsang-Gommern
  - 23, Würzburg
- Italy (2):
  - 29, Pavia
  - 34, Roma
- Poland (9):
  - 58, Bydgoszcz
  - 67, Elblag
  - 62, Lublin
  - 55, Poznan
  - 65, Poznan
  - 60, Sopot
  - 57, Szczecin
  - 69, Torun
  - 53, Warsaw

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects must have either failed to achieve remission in C87076 [NCT00674362] at Week 20 and/or Week 24 (CDAI >2.8), which was confirmed at Week 24, or must have achieved remission at Week 20, which was confirmed at Week 24, flared up between Week 24 and Week 52 and completed the entire C87076 study through Week 52.
Pre-assignment Details: Participant Flow refers to the Enrolled Set consisting of all subjects who gave informed consent.
Groups:
- Certolizumab Pegol: Certolizumab Pegol: 200 mg every two weeks
  Certolizumab Pegol 200 mg was administered every two weeks at the hospital by a nurse or at the patient's home done by patient (self-injection).
  Subjects who flared at Week 48 or Week 52 of feeder study C87076 [NCT00674362], received respectively once 400 mg Certolizumab Pegol or three times 400 mg Certolizumab Pegol at two weeks interval as part of an induction phase in the C87080 study. Thereafter the subject entered the C87080 study and was further treated with 200 mg Certolizumab Pegol every two weeks.
Period: Overall Study
Arm/Group | Certolizumab Pegol
Started | 131
Completed | 96
Not Completed | 35
Not completed — Adverse Event | 15
Not completed — Lack of Efficacy | 14
Not completed — Loss of efficacy | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: One subject did not receive treatment during C87080, so it is excluded from the Full Analysis Set (FAS) and Safety Set (SS).
  Full Analysis Set (FAS) consists of all subjects from the Enrolled Set who were dispensed medication.
  Safety Set is identical to the FAS.
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 113
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 25
Region of Enrollment [Number; unit: participants]
  Austria | 15
  France | 3
  Germany | 28
  Italy | 7
  Poland | 77

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Reporting At Least One Treatment-emergent Adverse Event (TEAE) During The Study Period
Description: A TEAE is defined as any untoward medical occurrence (eg, noxious or pathological changes) in a subject or clinical investigation subject compared with pre-existing conditions, that occurs during any phase of a clinical trial including Pretreatment, Run-In, Wash-Out, or Follow-Up Phases. A TEAE is defined as being independent of assumption of any causality (eg, to trial or concomitant medication, primary or concomitant disease, or trial design). TEAEs are all AEs in which the onset and time is after the first study drug administration in C87080, up to 70 days after the last injection.
Time Frame: From Entry Visit up to approximately 144 weeks
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
percentage of participants | 70.8

2. Primary Outcome: Percentage of Subjects With At Least One Treatment-emergent Serious Adverse Event (SAE) During The Study Period
Description: A Serious Adverse Event is any untoward medical occurrence that at any dose results in death, is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity is a congenital anomaly/birth defect.
Time Frame: From Entry Visit up to approximately 144 weeks
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
percentage of participants | 19.2

3. Secondary Outcome: Percentage of Subjects With DAS28[ESR] (Disease Activity Score 28 [Erythrocyte Sedimentation Rate]) Remission (DAS28[ESR] < 2.6) at Completion/Withdrawal Visit
Description: DAS28(ESR) is calculated using the tender joint count (TJC), swollen joint count (SJC) erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity. < 2.6 (Remission), > = 2.6 - < =3.2 Low, > 3.2 - < = 5.1 Moderate, > 5.1 High.
Time Frame: Completion/Withdrawal Visit (up to approximately Week 136)
Population: Of the 130 subjects in the Full Analysis Set, 114 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 114
percentage of participants | 34.2

4. Secondary Outcome: Percentage of Subjects With CDAI (Clinical Disease Activity Index) Remission (CDAI ≤2.8) at Completion/Withdrawal Visit
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined where a lower score indicates less disease activity. A lower CDAI score indicating improvement in activity and a higher score indicating a decline activity.
Time Frame: Completion/Withdrawal Visit (up to approximately Week 136)
Population: Of the 130 subjects in the Full Analysis Set, 122 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 122
percentage of participants | 27.9

5. Secondary Outcome: Percentage of Subjects With SDAI (Simplified Disease Activity Index) Remission (SDAI ≤3.3) at Completion/Withdrawal Visit
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined where a lower score indicates less disease activity. <= 3.3 (Remission), >3.3 - <= 11 Low, > 11 - <= 26 Moderate, > 26 High.
Time Frame: Completion/Withdrawal Visit (up to approximately Week 136)
Population: Of the 130 subjects in the Full Analysis Set, 120 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 120
percentage of participants | 25.8

6. Secondary Outcome: Percentage of Subjects With ACR20 (American College of Rheumatology 20 % Improvement) Response at Completion/Withdrawal Visit
Description: ACR20 response is defined for subjects with at least 20 % improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire- Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity, 5) Physician's Global Assessment of Disease Activity.
Time Frame: Baseline in the feeder study (C87076 [NCT00674362]) to Completion/Withdrawal Visit in the extension study (up to approximately Week 136)
Population: Of the 130 subjects in the Full Analysis Set, 124 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 124
percentage of participants | 57.3

7. Secondary Outcome: Percentage of Subjects With ACR50 (American College of Rheumatology 50 % Improvement) Response at Completion/Withdrawal Visit
Description: ACR50 response is defined for subjects with at least 50 % improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire- Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity, 5) Physician's Global Assessment of Disease Activity.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 124
percentage of participants | 35.5

8. Secondary Outcome: Percentage of Subjects With ACR70 (American College of Rheumatology 70 % Improvement) Response at Completion/Withdrawal Visit
Description: ACR70 response is defined for subjects with at least 70 % improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire- Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity, 5) Physician's Global Assessment of Disease Activity.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 124
percentage of participants | 15.3

9. Secondary Outcome: Change From Baseline in HAQ-DI (Health Assessment Questionnaire-Disability Index) at Completion/Withdrawal Visit
Description: HAQ-DI is derived based on the mean of individual scores in 8 categories of daily living activities (using 20 questions). Each question is scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). Thus, the mean also has a range from 0-3. Change from Baseline is computed as the value at Completion/Withdrawal minus the Baseline value. A negative value in change from Baseline indicates an improvement.
Time Frame: as for outcome 6
Population: Of the 130 subjects in the Full Analysis Set, 119 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 119
units on a scale | -0.36 (0.55)

10. Secondary Outcome: Change From Baseline in PtAAP (Patient's Assessment of Arthritis Pain) at Completion/Withdrawal Visit
Description: Change from Baseline in Patient's Assessment of Arthritis Pain - Visual Analog Scale (VAS) (0 to 100 mm visual analog scale, 0 being no pain and 100 being most severe pain) is computed as the value at Completion/Withdrawal minus the Baseline value. A negative value in change from Baseline indicates an improvement.
Time Frame: as for outcome 6
Population: Of the 130 subjects in the Full Analysis Set, 102 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 102
units on a scale | -15.90 (23.72)

11. Secondary Outcome: Change From Baseline in FAS (Fatigue Assessment Scale) at Completion/Withdrawal Visit
Description: Change from Baseline in Fatigue Assessment Scale (0 to 10, 0 is "No Fatigue" and 10 is "Fatigue as bad as you can imagine") is computed as the value at Completion/Withdrawal minus the Baseline value. A negative value in change from Baseline indicates an improvement.
Time Frame: as for outcome 6
Population: Of the 130 subjects in the Full Analysis Set, 117 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 117
units on a scale | -1.23 (2.43)

12. Secondary Outcome: Change From Baseline in PtGADA (Patient's Global Assessment of Disease Activity) at Completion/Withdrawal Visit
Description: Change from Baseline in Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS) (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as the value at Completion/Withdrawal minus the Baseline value. A negative value in change from Baseline indicates an improvement.
Time Frame: Baseline in the feeder study (C87076 [NCT00674362]) to Completion/Withdrawal Visit in the extension study (up to Week approximately 136)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 119
units on a scale | -13.18 (23.73)

13. Secondary Outcome: Geometric Mean of Plasma Concentration of Certolizumab Pegol at Week 24 Visit
Description: Plasma Samples for determination of Certolizumab Pegol were taken prior to Certolizumab Pegol administration. Values below the limit of quantification of 0.41 μg/mL will be set to half the limit of quantification for the summaries (0.205 μg/mL).
Time Frame: Week 24
Population: Of the 130 subjects in the Safety Set, 89 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 89
μg/mL | 17.091 [14.981 to 19.499]

14. Secondary Outcome: Percentage of Subjects With Positive Anti-Certolizumab Pegol (CZP) Antibody Status at Any Time From Baseline of the Feeder Study C87076 to the Completion/Withdrawal Visit of the Extension Study
Description: Antibody positive is defined as Anti-CZP antibody levels > 2.4 units/mL at any visit.
Time Frame: as for outcome 6
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
percentage of participants | 10.0

15. Secondary Outcome: Percentage of Subjects Willing to Self-inject at Week 0
Description: The percentage of subjects willing to self-inject at Week 0 will be presented using the Full Analysis Set.
Time Frame: Week 0 of this study (C87080 [NCT00843778])
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
percentage of participants | 69.2

16. Secondary Outcome: Mean PRE-Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 0
Description: The three domains of the PRE SIAQ are feelings about injections, self-confidence, and satisfaction with self-injection. The SIAQ items are scored on a semantic Likert-type scale where lower numbers indicate a worse experience. Domain scores range from 0 to 10. Subjects self-injecting completed this pre-self-injection questionnaire. The PRE-SIAQ is taken before the subject's first injection.
Time Frame: Week 0 of this study (C87080 [NCT00843778])
Population: Of the 130 subjects in the Full Analysis Set, 66 subjects are included in the analysis of each subscale measure, based upon the number of subjects self-injecting at the visit, with the available subscale score at the visit. For each subscale of the questionnaire, N, Mean and SD are presented for non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
units on a scale
  Feelings about injections (N = 66) | 7.929 (1.979)
  Self-confidence (N = 66) | 5.922 (2.174)
  Satisfaction with self-injection (N = 66) | 7.462 (2.033)

17. Secondary Outcome: Mean POST-Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 0
Description: The six domains of the POST SIAQ are feelings about injections, self-image, self-confidence, injection-site reactions, ease of use, and satisfaction with self-injection. The SIAQ items are scored on a semantic Likert-type scale where lower numbers indicate a worse experience. Domain scores range from 0 to 10. Subjects self-injecting at this visit completed this SIAQ questionnaire. The POST-SIAQ is taken after the injection at that visit.
Time Frame: Week 0 of this study (C87080 [NCT00843778])
Population: Of the 130 subjects in the Full Analysis Set, 65 or 66 subjects are included in the analysis of each subscale measure, based upon the number of subjects self-injecting at the visit, with the available subscale score at the visit. For each subscale of the questionnaire, N, Mean and SD are presented for non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
units on a scale
  Feelings about injections (N = 66) | 8.093 (1.853)
  Self-image (N = 66) | 8.295 (2.243)
  Self-confidence (N = 66) | 6.881 (1.839)
  Injection-site reactions (N = 66) | 9.206 (1.158)
  Ease of use (N = 65) | 7.376 (1.579)
  Satisfaction with self-injection (N = 65) | 6.994 (0.909)

18. Secondary Outcome: Mean POST-Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 2
Description: as for outcome 17
Time Frame: Week 2
Population: Of the 130 subjects in the Full Analysis Set, 80 or 81subjects are included in the analysis of each subscale measure, based upon the number of subjects self-injecting at the visit, with the available subscale score at the visit. For each subscale of the questionnaire, N, Mean and SD are presented for non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
units on a scale
  Feelings about injections (N = 81) | 8.076 (1.979)
  Self-image (N = 80) | 8.313 (2.019)
  Self-confidence (N = 80) | 6.719 (1.905)
  Injection-site reactions (N = 81) | 8.984 (1.376)
  Ease of use (N = 80) | 7.250 (1.790)
  Satisfaction with self-injection (N =81) | 6.847 (1.184)

19. Secondary Outcome: Mean POST-Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 4
Description: as for outcome 17
Time Frame: Week 4
Population: Of the 130 subjects in the Full Analysis Set, 82 or 83 subjects are included in the analysis of each subscale measure, based upon the number of subjects self-injecting at the visit, with the available subscale score at the visit. For each subscale of the questionnaire, N, Mean and SD are presented for non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
units on a scale
  Feelings about injections (N = 83) | 8.213 (1.785)
  Self-image (N = 83) | 8.434 (1.941)
  Self-confidence (N = 83) | 6.847 (1.707)
  Injection-site reactions (N = 82) | 9.013 (1.360)
  Ease of use (N = 82) | 7.512 (1.607)
  Satisfaction with self-injection (N = 83) | 6.995 (1.100)

20. Secondary Outcome: Mean POST-Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 6
Description: as for outcome 17
Time Frame: Week 6
Population: Of the 130 subjects in the Full Analysis Set, 66, 67 or 68 subjects are included in the analysis of each subscale measure, based upon the number of subjects self-injecting at the visit, with the available subscale score at the visit. For each subscale of the questionnaire, N, Mean and SD are presented for non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
units on a scale
  Feelings about injections (N = 68) | 8.407 (1.732)
  Self-image (N = 67) | 8.545 (1.854)
  Self-confidence (N = 68) | 6.777 (2.225)
  Injection-site reactions (N = 67) | 9.025 (1.357)
  Ease of use (N = 66) | 7.982 (1.308)
  Satisfaction with self-injection (N = 68) | 7.068 (1.042)

21. Secondary Outcome: Mean POST-Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 8
Description: as for outcome 17
Time Frame: Week 8
Population: Of the 130 subjects in the Full Analysis Set, 78, 79 or 80 subjects are included in the analysis of each subscale measure, based upon the number of subjects self-injecting at the visit, with the available subscale score at the visit. For each subscale of the questionnaire, N, Mean and SD are presented for non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
units on a scale
  Feelings about injections (N = 80) | 8.458 (1.635)
  Self-image (N = 80) | 8.563 (1.769)
  Self-confidence (N = 80) | 6.854 (1.842)
  Injection-site reactions (N = 78) | 9.214 (1.144)
  Ease of use (N = 79) | 7.585 (1.401)
  Satisfaction with self-injection (N = 80) | 7.112 (0.971)

22. Secondary Outcome: Mean POST-Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 10
Description: as for outcome 17
Time Frame: Week 10
Population: Of the 130 subjects in the Full Analysis Set, 72, 73 or 74 subjects are included in the analysis of each subscale measure, based upon the number of subjects self-injecting at the visit, with the available subscale score at the visit. For each subscale of the questionnaire, N, Mean and SD are presented for non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
units on a scale
  Feelings about injections (N = 74) | 8.446 (1.730)
  Self-image (N = 72) | 8.472 (1.948)
  Self-confidence (N = 74) | 7.050 (1.852)
  Injection-site reactions (N = 73) | 8.908 (1.459)
  Ease of use (N = 73) | 7.792 (1.488)
  Satisfaction with self-injection (N = 73) | 7.105 (0.876)

23. Secondary Outcome: Mean POST-Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 12
Description: as for outcome 17
Time Frame: Week 12
Population: Of the 130 subjects in the Full Analysis Set, 74 or 75 subjects are included in the analysis of each subscale measure, based upon the number of subjects self-injecting at the visit, with the available subscale score at the visit. For each subscale of the questionnaire, N, Mean and SD are presented for non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 130
units on a scale
  Feelings about injections (N = 75) | 8.467 (1.673)
  Self-image (N = 74) | 8.446 (2.057)
  Self-confidence (N = 75) | 7.122 (1.803)
  Injection-site reactions (N = 75) | 9.038 (1.513)
  Ease of use (N = 74) | 7.973 (1.335)
  Satisfaction with self-injection (N = 75) | 7.127 (0.975)

24. Secondary Outcome: Mean Injection Site Reaction Questionnaire (ISRQ) Score at Week 0
Description: The ISRQ is scored on a semantic Likert-type scale where lower numbers indicate a worse experience. Scores range from 0 to 10. Subjects receiving hospital nurse injection at this visit completed the ISRQ questionnaire.
Time Frame: Week 0
Population: Of the 130 subjects in the Full Analysis Set, 31 subjects are included in the analysis of this outcome measure, based upon the number of subjects receiving hospital nurse injection at this visit, with an available assessment score at the visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 31
units on a scale | 9.588 (0.471)

25. Secondary Outcome: Mean Injection Site Reaction Questionnaire (ISRQ) Score at Week 2
Description: as for outcome 24
Time Frame: Week 2
Population: Of the 130 subjects in the Full Analysis Set, 36 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 36
units on a scale | 9.688 (0.448)

26. Secondary Outcome: Mean Injection Site Reaction Questionnaire (ISRQ) Score at Week 4
Description: as for outcome 24
Time Frame: Week 4
Population: Of the 130 subjects in the Full Analysis Set, 35 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 35
units on a scale | 9.804 (0.340)

27. Secondary Outcome: Mean Injection Site Reaction Questionnaire (ISRQ) Score at Week 6
Description: as for outcome 24
Time Frame: Week 6
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 36
units on a scale | 9.705 (0.388)

28. Secondary Outcome: Mean Injection Site Reaction Questionnaire (ISRQ) Score at Week 8
Description: as for outcome 24
Time Frame: Week 8
Population: Of the 130 subjects in the Full Analysis Set, 34 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 34
units on a scale | 9.634 (0.423)

29. Secondary Outcome: Mean Injection Site Reaction Questionnaire (ISRQ) Score at Week 10
Description: as for outcome 24
Time Frame: Week 10
Population: Of the 130 subjects in the Full Analysis Set, 37 subjects are included in the analysis of this outcome measure, based upon the number of subjects with an available assessment at the visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 37
units on a scale | 9.771 (0.335)

30. Secondary Outcome: Mean Injection Site Reaction Questionnaire (ISRQ) Score at Week 12
Description: as for outcome 24
Time Frame: Week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 37
units on a scale | 9.611 (0.652)

ADVERSE EVENTS:
Time Frame: From entry visit up to approximately 144 weeks
Description: Adverse Events refer to the Safety Set consisting of all enrolled subjects who were dispensed medication.
Groups:
- Certolizumab Pegol: Certolizumab Pegol: 200 mg every two weeks
  Certolizumab Pegol 200 mg was administered every two weeks at the hospital by a nurse or at the patient's home done by patient (self-injection).
  Subjects who flared at Week 48 or Week 52 of feeder study C87076 [NCT00674362], will receive respectively once 400 mg Certolizumab Pegol or three times 400 mg Certolizumab Pegol at two weeks interval as part of an induction phase in the C87080 study. Thereafter the subject enters the C87080 study and will be further treated with 200 mg Certolizumab Pegol every two weeks.
Arm/Group | Certolizumab Pegol
Serious Adverse Events (participants affected / at risk) | 25/130
Other Adverse Events (participants affected / at risk) | 35/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=130)
Myocardial Ischaemia (Cardiac disorders) | 2 (2)
Goitre (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Hepatitis Toxic (Hepatobiliary disorders) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
Bronchitis Acute (Infections and infestations) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 1 (1)
Wound Infection Staphylococcal (Infections and infestations) | 1 (1)
Lymph Node Tuberculosis (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 1 (1)
Silicosis (Injury, poisoning and procedural complications) | 1 (1)
Patella Fracture (Injury, poisoning and procedural complications) | 1 (1)
Knee Deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Destruction (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Instability (Musculoskeletal and connective tissue disorders) | 1 (2)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Colpocele (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hip Arthroplasty (Surgical and medical procedures) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Certolizumab Pegol (N=130)
Diarrhoea (Gastrointestinal disorders) | 8
Nasopharyngitis (Infections and infestations) | 8
Pharyngitis (Infections and infestations) | 8
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days